CLINICAL TRIAL: NCT05623384
Title: Effect of Ultrasound-guided Stellate Ganglion Block Combined With Facial Nerve and Glossopharyngeal Nerve Block on the Treatment of Sudden Deafness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhuan Zhang (Other)
Responsible Party: Sponsor-Investigator, Zhuan Zhang, Clinical Professor, Yangzhou University
Organization: Yangzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20221031
Record Dates: First submitted 2022-11-13; First posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Sudden Deafness
Keywords: Sudden deafness; Stellate Ganglion Block; Facial nerve block; Glossopharyngeal nerve block
MeSH Terms: conditions — Hearing Loss, Sudden | interventions — mecobalamin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stellate ganglion block combined with facial and glossopharyngeal nerve block group (Experimental)
  Interventions: Procedure: Stellate ganglion block; Procedure: Facial and glossopharyngeal nerve blocks; Drug: Mecobalamin Tablets
- Stellate ganglion block group (Experimental)
  Interventions: Procedure: Stellate ganglion block; Drug: Mecobalamin Tablets
- Control group (Other)
  Interventions: Drug: Mecobalamin Tablets

INTERVENTIONS:
Procedure: Stellate ganglion block — A cross-sectional scan with a high-frequency line array probe reveals the pre-C6 transverse nodule or C7 transverse process, and the structures of the thyroid, carotid sheath, vertebral artery, inferior thyroid artery, trachea, and esophagus are identified by observation. The carotid sheath is pushed out as far as possible laterally, the needle is inserted in the paratracheal sulcus, and the tip of the needle is passed through the lateral border of the thyroid into the deep anterior fascial surface of the long cervical muscle.After backdrawing no blood, cerebrospinal fluid or gas, 5 ml of lidocaine was injected.（lidocaine 80mg；Physiological saline 1ml）
  Arms: Stellate ganglion block combined with facial and glossopharyngeal nerve block group; Stellate ganglion block group
Procedure: Facial and glossopharyngeal nerve blocks — The operator touches the position of the mastoid process and needles vertically at the front of the mastoid process directly below the external auditory canal. When the surface of the mastoid is touched, the needle is adjusted to pass through the front of the mastoid and then slowly needled for about 1 cm, and when the patient develops swelling and pain, 3 ml of the drug is injected. then the needle is slowly needled backward for about 1 cm, and when the patient develops swelling and pain, 2 ml of the drug is injected. （mecobalamin injection 1mg；lidocaine 20mg； dexamethasone 10mg ；Physiological saline 2ml）
  Arms: Stellate ganglion block combined with facial and glossopharyngeal nerve block group
Drug: Mecobalamin Tablets — oral Mecobalamin Tablets tid-8

SUMMARY:
Sudden deafness is a sudden, unexplained sensorineural hearing loss of ≥20 dBHL in at least two adjacent frequencies within 72 h. It may be accompanied by tinnitus, a sense of ear congestion, vertigo and other Symptoms.Stellate ganglion block increases the blood flow and blood velocity in the inner ear, keeping the body's vegetative, endocrine and immune functions normal.The branches of the facial and linguopharyngeal nerves are connected to the inner ear, and local injection can nourish the nerves and improve local circulation.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for sudden deafness established by the Editorial Board of the Chinese Journal of Otolaryngology, Head and Neck Surgery and the Chinese Society of Otolaryngology, Head and Neck Surgery
* Age 18 to 80 years
* ASA classification Ⅰ~Ⅲ grade

Exclusion Criteria:

* Acoustic conductance test, vestibular function test, cranial MRI, etc. suggest organic disease
* People with coagulation disorders or on anticoagulation therapy
* Infection at the puncture site
* Severe systemic diseases that cannot cooperate with treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Mean Hearing Threshold (PTA) | Baseline (Before treatment)，1 month and 2 months after treatment
  The average of hearing thresholds at six frequencies (250, 500, 1000, 2000, 4000, and 8000 Hz) was recorded as the mean hearing threshold (PTA).

CONTACTS AND LOCATIONS:
Overall Officials: zhuan zhang, professor, Principal Investigator — The Affiliated Hospital of Yangzhou University
Locations (1):
- the Affiliated Hospital of Yangzhou University, Yangzhou, Jiangsu, China